CLINICAL TRIAL: NCT07262372
Title: Supervision Strategy for Substance Use Disorder Treatment Programs: A Pilot Study
Brief Title: Supervision in Substance Use Disorder Treatment Programs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Chestnut Health Systems (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 297361; R34DA060419 (NIH)
Record Dates: First submitted 2025-11-12; First posted 2025-12-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Self Efficacy; Burnout, Professional; Substance Use Disorders; Supervision
Keywords: supervision; substance use disorder treatment facility; organizational context; counselor burnout; counselor self-efficacy
MeSH Terms: conditions — Burnout, Professional; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: One arm pilot/feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supervision arm (Experimental): Supervisors will be trained and coached in a new supervision strategy (FOCUS)
  Interventions: Other: FOCUS supervision strategy

INTERVENTIONS:
Other: FOCUS supervision strategy — The FOCUS supervision strategy provides a strenghts-based model for supervision. It is built around three core components: (1) Five pillars for effective supervision interactions, (2) practical skills that operationalize these principles, and (3) a set of experiential activities that provide foundational learnings for staff to practice the skills around real-life situations (from which future client-specific interventions can be built). In this study, FOCUS is being tailored for SUD treatment settings.

SUMMARY:
Substance use disorders such as opioid addiction affect millions of adults in the United States each year, but the delivery of high-quality, effective addiction services is disrupted by organizational issues such as counselor burnout and turnover. Clinical supervisors are essential for supporting counselors in specialty addiction treatment programs, but few supervisors receive supervision-focused training. This project seeks to develop and pilot an evidence-based supervision strategy that has a high potential to enhance supervision and result in improved counselors' well-being and performance and, in turn, to improve client outcomes.

DETAILED DESCRIPTION:
Substance use disorders (SUDs) such as addiction to opioids, methamphetamines and alcohol are a significant burden in the US, affecting almost 50 million individuals annually. Community specialty SUD treatment programs ("SUD programs") are a key type of SUD providers and while effective treatments for SUD exist, significant issues in the organization and delivery of SUD programs (e.g., burnout, turnover) undermine the delivery of high-quality services. Clinical supervisors are centrally positioned to support SUD counselors (frontline clinical providers) and ensure high service quality. For clinical supervisors to effectively support counselors, they need evidence-based supervision strategies. Currently, supervisors in community SUD programs receive very little training, support, and direction for supervision, and thus their supervision practices are highly variable, raising concern about the effectiveness of clinical supervision as currently provided in these programs. Evidence-based supervision strategies can help fill the gap, and evidence from child welfare settings shows they improve leadership, climate, and client outcomes. Based on our preliminary formative work with SUD providers in Arkansas, a reinforcement-based supervision strategy developed for counselors was deemed acceptable and feasible in SUD programs, and had high perceived potential to improve supervision quality, counselor well-being and performance, and client outcomes. Participants thought the structure and content of the strategy were a good fit for SUD settings. However, for a supervision strategy to be supportive of the work they do, it needs to be developed to reflect the language, case examples, and organizational factors relevant to the SUD settings. The goals of our study are to iteratively develop and refine a supervision strategy for SUD settings, and to pilot it in residential treatment programs using quality improvement and implementation science tools and approaches. Aim 1 involves leveraging previous experience developing supervision strategies and partnering with SUD providers to develop and refine the supervision strategy for SUD. Using the Evidence-Based Quality Improvement (EBQI) process, we will engage SUD partners in a series of collaborative meetings to review and discuss the supervision strategy and related study materials, and to make key decisions. The output of this work will be a refined and optimized SUD supervision strategy. Aim 2 involves conducting two pilot cycles with supervisors and counselors in a sample of SUD residential treatment programs to assess the feasibility and acceptability of the supervision strategy, examine its impact on key organizational, counselor, and client outcomes, and to document barriers and facilitators for its implementation and sustained use in routine practice. This study will provide key information to inform planning and design of a future fully powered study to assess the effectiveness of the new supervision strategy in a large sample of SUD programs.

ELIGIBILITY:
Inclusion Criteria:

* Serves as a supervisor (i.e., oversee work of counselors) or counselor (i.e., directly work with clients) at a substance use treatment facility/program
* Program/facility provides residential services

Exclusion Criteria:

* Supervisors contracted (not employed) by the facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Counselor self-efficacy | Every 6 months for 2 years
  Self-reported survey response at the counselor level (Efficacy subscale on TCU ORC; 1-5 Likert scale, higher scores are better; Lehman WEK, Greener JM, Simpson DD. Assessing organizational readiness for change. J Subst Abuse Treat. 2002;22(4):197-209. doi: 10.1016/S0740-5472(02)00233-7.)

SECONDARY OUTCOMES:
Supervisor fidelity to FOCUS | Monthly, 2 years
  Expert rated fidelity to FOCUS at the supervisor level (measure to be developed as part of the study)
FOCUS acceptability | Every 6 months, for 2 years
  Supervisor perceptions of acceptability (satisfaction, appeal) of FOCUS and related materials (Acceptability of Intervention Measure [AIM], 1-5 Likert scale, higher scores are better; Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Science. 2017;12:1-12. doi: 10.1186/s13012-017-0635-3.)
FOCUS feasibility | Every 6 months, for 2 years
  Supervisor perceptions of feasibility (ease of use, "do-ability") of FOCUS and related materials (Feasibility of Intervention Measure [FIM], 1-5 Likert scale, higher scores are better; Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. Implementation Science. 2017;12:1-12. doi: 10.1186/s13012-017-0635-3.)
Leadership - implementation leadership | Every 6 months, for 2 years
  Counselor perceptions of supervisors' support for ESTs (Implementation Leadership Scale [ILS], 1-5 Likert scale, higher scores are better; Aarons GA, Ehrhart MG, Torres EM, Finn NK, Roesch SC. Validation of the implementation leadership scale (ILS) in substance use disorder treatment organizations. J Subst Abuse Treat. 2016;68:31-35. doi: 10.1016/j.jsat.2016.05.004.)
Leadership - clinical supervision | Every 6 months, for 2 years
  Counselor perceptions of supervisor instrumental assistance (Clinical Supervision, 1-5 Likert scale, higher scores are better; Knudsen HK, Ducharme LJ, Roman PM. Clinical supervision, emotional exhaustion, and turnover intention: A study of substance abuse treatment counselors in the clinical trials network of the national institute on drug abuse. J Subst Abuse Treat. 2008;35(4):387-395. doi: 10.1016/j.jsat.2008.02.003.)
Organizational Social Context - implementation climate | Every 6 months, for 2 years
  Supervisor and counselor shared perceptions of organizational expectations of, and support and reward for EST use (Implementation Climate Scale [ICS], 1-5 Likert scale, higher scores are better; Ehrhart MG, Torres EM, Hwang J, Sklar M, Aarons GA. Validation of the implementation climate scale (ICS) in substance use disorder treatment organizations. Substance abuse treatment, prevention, and policy. 2019;14(1):1-10. doi: 10.1186/s13011-019-0222-5.)
Organizational Social Context - organizational climate | Every 6 months, for 2 years
  Supervisor and counselor shared perceptions of organizational environment (Mission, Cohesion, and Stress subscales from TCU ORC; and Effort subscale from the Patterson Organizational Climate Measure; 1-5 Likert scale, higher scores are better; responses will be aggregated across subscales for primary analyses; Lehman WEK, Greener JM, Simpson DD. Assessing organizational readiness for change. J Subst Abuse Treat. 2002;22(4):197-209. and Patterson MG, West MA, Shackleton VJ, et al. Validating the organizational climate measure: Links to managerial practices, productivity and innovation. J Organ Behav. 2005;26(4):379-408. doi: 10.1002/job.312.)
Counselor functioning - burnout | Every 6 months, for 2 years
  Counselor perceptions of being overextended and depleted of emotional and physical resources (Emotional Exhaustion on Maslach Burnout Inventory; 1-5 Likert scale, lower scores are better; Maslach C, Jackson SE. The measurement of experienced burnout. J Organ Behav. 1981;2(2):99-113. doi: 10.1002/job.4030020205.)
Counselor performance | Every 6 months, for 2 years
  Supervisor ratings of counselor performance (based on annual performance evaluations in use at the facilities)
Organizational performance/outcomes - turnover | Every 6 months, for 2 years
  Objective measures of employee turnover rate (at program level)
Organizational performance/outcomes - client treatment completion | Every 6 months, for 2 years
  Objective measures of client treatment completion rate (at program level)
Organizational performance/outcomes - client satisfaction | Every 6 months, for 2 years
  Client-reported satisfaction levels (at program level; as routinely collected by programs)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data will include observational data on supervisor fidelity (expert ratings); survey data on leadership, organizational social context, and counselor functioning (self-reported by counselors and/or supervisors); and interview data with leadership, supervisors, and counselors based on semi-structured interview guides informed by the study conceptual model and implementation science framework.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Estimated in 2027 (at study conclusion and submission of manuscripts); We will archive our data in NAHDAP (https://www.icpsr.umich.edu/web/pages/NAHDAP/) following the Restricted-Use Data Deposit and Dissemination Procedures.
Access Criteria: We will archive our data in NAHDAP following Restricted-Use Data Deposit and Dissemination Procedures.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/